CLINICAL TRIAL: NCT05781594
Title: Family Cohort Study on Primary Osteoporosis With Kidney-yang Deficiency Syndrome
Brief Title: Family Cohort Study on Primary Osteoporosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: ShanghaiUTCM20230201
Record Dates: First submitted 2023-02-05; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Family Genetic Characteristics of Osteoporosis
Keywords: Osteoporosis families; Kidney-yang deficiency; Genetic correlation of disease; Bone density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Serum, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bone metabolism and genetic characteristics of osteoporosis pedigree with kidney-yang deficiency

DETAILED DESCRIPTION:
Families with or without osteoporosis of kidney-yang deficiency type will be included and compared with each other. Their genetic characteristics, bone changes, and TCM constitution are the focus of research.

ELIGIBILITY:
Inclusion Criteria:

* Be able to cooperate with inspection.There is blood relationship between the members of the enrolled family.

Exclusion Criteria:

* Unable to cooperate with inspection.There is not blood relationship between the members of the enrolled family.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: member of family
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
changes in bone mineral density from baseline to 5 years after enrollment | at enrollment
  lumbar (L1-4 as well as total) and hip bone mineral density will be recorded by dual energy X-ray absorptiometry
changes in bone mineral density from baseline to 5 years after enrollment | 5 years after enrollment
  lumbar (L1-4 as well as total) and hip bone mineral density will be recorded by dual energy X-ray absorptiometry
Physical phenotype of traditional Chinese medicine | at enrollment
  Occurrence of kidney yang deficiency
Physical phenotype of traditional Chinese medicine | 5 years after enrollment
  Occurrence of kidney yang deficiency
Understand the general situation through the questionnaire | at enrollment
  Including age（year）, sex（man,wowan）, height(cm), weight(kg), menstrual period,history of smoking and drinking, living habits, fracture history and risk assessment, skeletal muscle assessment, living environment, Chinese medicine constitution, etc
Understand the general situation through the questionnaire | 5 years after enrollment
  Including age（year）, sex（man,wowan）, height(cm), weight(kg), menstrual period,history of smoking and drinking, living habits, fracture history and risk assessment, skeletal muscle assessment, living environment, Chinese medicine constitution, etc

SECONDARY OUTCOMES:
Osteocalcin | at enrollment
  serum osteocalcin
procollagen type I N-terminal propeptide | at enrollment
  serum procollagen type I N-terminal propeptide (PINP)
Bone alkaline phosphatase | at enrollment
  serum bone alkaline phosphatase (BALP)
β-crosslaps | at enrollment
  serum β-crosslaps (β-CTX)
Ca | at enrollment
  serum Ca
P | at enrollment
  serum P
Mg | at enrollment
  serum Mg
Fibroblast growth factor | at enrollment
  serum fibroblast growth factor (FGF)23
Parathormone | at enrollment
  serum parathormone (PTH)
25(OH) vitamin D | at enrollment
  serum total 25(OH) vitamin D
Osteocalcin | 5 years after enrollment
  serum osteocalcin
Procollagen type I N-terminal propeptide | 5 years after enrollment
  serum procollagen type I N-terminal propeptide (PINP)
Bone alkaline phosphatase | 5 years after enrollment
  serum bone alkaline phosphatase (BALP)
β-crosslaps | 5 years after enrollment
  serum β-crosslaps (β-CTX)
Ca | 5 years after enrollment
  serum Ca
P | 5 years after enrollment
  serum P
Mg | 5 years after enrollment
  serum Mg
Fibroblast growth factor | 5 years after enrollment
  serum fibroblast growth factor (FGF)23
Parathormone | 5 years after enrollment
  serum parathormone (PTH)
25(OH) vitamin D | 5 years after enrollment
  serum total 25(OH) vitamin D
Gene testing(BGIseq T5,WGS) | at enrollment
  Carry out whole-gene testing on the samples with obvious family heritability of osteoporosis, and analyze the differences at the gene level through sequencing compared with the control group
Gene testing(BGIseq T5,WGS) | 5 years after enrollment
  Carry out whole-gene testing on the samples with obvious family heritability of osteoporosis, and analyze the differences at the gene level through sequencing compared with the control group

CONTACTS AND LOCATIONS:
Overall Officials: Yongjun Wang, Study Chair — Shanhgai University of TCM; Chuanglong Xu, Study Director — Ningxia Chinese medicine Rearch Center; Zhangyu Liao, Study Director — Nankang Traditional Chinese Medicine Hospital
Locations (3):
- China (3):
  - Nankang Traditional Chinese Medicine Hospital, Gannan, Jiangxi
  - Ningxia Chinese medicine Rearch Center, Yinchuan, Ningxia
  - Longhua Hospital, Shanghai University of TCM, Shanghai

IPD SHARING:
Plan to Share IPD: No